CLINICAL TRIAL: NCT04373317
Title: CSP #2015 - Multicenter, Randomized, Double-blind Comparator Study of Antipsychotics Pimavanserin and Quetiapine for Parkinson''s Disease Psychosis (C-SAPP)
Brief Title: Pimavanserin vs. Quetiapine for Treatment of Parkinson's Psychosis
Acronym: C-SAPP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Parkinson's Disease Psychosis
Keywords: Pimavanserin; Quetiapine
MeSH Terms: interventions — pimavanserin; Quetiapine Fumarate

STUDY DESIGN:
Intervention Model Description: Two active treatments will be administered in this RCT, with 1:1 treatment assignment to either quetiapine or pimavanserin. Both active treatments are FDA-approved antipsychotics.
Who Masked: Participant, Care Provider, Investigator
Masking Description: In order to facilitate titrations, study drug will be provided in blister cards with a sufficient number of over-encapsulated drug to bridge participants to their next titration step. Each blister card will contain a one-week supply of study drug. Because dosing will be nightly, and the study will use a combination of quetiapine strengths for all protocol-specified quetiapine doses, participants in both treatment groups will take two identical capsules both of which containing the protocol-specified nightly dose. For example, if a participant is randomized to quetiapine and is up-titrated from 50 to 100 mg ER, this participant will take 2 identical capsules, each containing 50 mg of ER quetiapine. Similarly, participants randomized to pimavanserin will take two capsules every night, one containing a placebo capsule, and the other containing 34 mg of pimavanserin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pimavanserin 34mg (Active Comparator): Participants assigned to pimavanserin will receive 34mg (equivalent to 40 mg pimavanserin tartrate) daily without titration; however, because pimavanserin is blinded to quetiapine, participants will undergo sham titration based on tolerability.
  Interventions: Drug: Pimavanserin
- Quetiapine (Active Comparator): Participants assigned to Quetiapine will be titrated from 25mg/day to a maximum of 200mg/day based on tolerability. During the 8-week treatment phase, there is a maximum of 6 weeks for titration.
  Titration Schedule
  Visit/call Quetiapine Dose (Flexible)Quetiapine Notes Baseline visit (Visit 00)25 mg IR QHSAll participants must be up-titrated to at least 50 mg/day at week 1 Week 1 call (Visit 01)50 mg XR QHS Up-titration Week 3 visit (Visit 03)100 mg XR QHS (requiring two 50-mg quetiapine XR capsules)Up- or down-titration as appropriate based on psychosis symptoms and tolerability Week 5 visit (Visit 05)150 mg quetiapine XR QHS Up- or down-titration as appropriate based on psychosis symptoms and tolerability Week 6 call (Visit 06)200 mg quetiapine XR QHS Up- or down-titration as appropriate based on psychosis symptoms and tolerability
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Pimavanserin — Fixed-dose Pimavanserin - Pimavanserin is a new antipsychotic agent, and pure 5HT-2A inverse agonist, that was approved by the FDA recently (2016) for the treatment of PDP. It is the only FDA-approved medication for PDP, but is still not the first-line AP used in PD. All participants assigned to pimavanserin will receive the FDA-approved dose of 34 mg (equivalent to 40 mg pimavanserin tartrate) daily without titration up or down; however, because pimavanserin is blinded to quetiapine, participants will undergo sham titration based on tolerability (i.e., overall adverse event profile) and efficacy (i.e., improvement in severity of psychosis).
  Arms: Pimavanserin 34mg
Drug: Quetiapine — Flexible-dose Quetiapine - Quetiapine, which is a mixed serotonin and dopamine receptor antagonist, is by far the most commonly used AP for PDP. However, scientific evidence for the efficacy of quetiapine in PDP is almost non-existent as most of the studies were underpowered, had high drop-out rates, and possibly underdosed quetiapine. Quetiapine immediate and extended release will be titrated as shown:
  Baseline visit Quetiapine: 25 mg IR QHS, All participants must be up-titrated to 50 mg/day
  Week 1 call Quetiapine: 50 mg XR QHS, Up-titration to 50 mg
  Week 3 visit Quetiapine: 100 mg XR QHS, Up-titration as appropriate
  Week 5 visit Quetiapine: 150 mg XR QHS, Up- or down-titration as appropriate
  Week 6 call Quetiapine: 200 mg XR QHS, Up- or down-titration as appropriate
  Arms: Quetiapine

SUMMARY:
Patients with Parkinson's disease (PD) sometimes experience symptoms affecting their movement, such as slowness, tremor, stiffness, and balance or walking problems. Many patients also have other symptoms not related to movement, called non-motor symptoms, which may affect one's mood or emotions, memory or thinking, or cause one to see or hear things that aren't real (hallucinations) or believe things that aren't true (delusions). Hallucinations or delusions, together called psychosis, occur in up to 60% of PD patients at some point in time. Parkinson's disease psychosis can sometimes be associated with decreased quality of life, increased nursing home placement, increased rate of death, and greater caregiver burden. There are approximately 50,000 Veterans with Parkinson's disease receiving care in the VA, and up to 30,000 (60%) of them will experience psychosis at some point in time.

Quetiapine is an antipsychotic drug approved by the Food and Drug Administration (FDA) that is the most commonly used medication to treat PD psychosis, but more studies are needed to determine if it works for this condition and is also well tolerated and safe. Pimavanserin is a newer antipsychotic drug approved by the Food and Drug Administration (FDA) specifically to treat PD psychosis, but more studies are needed to determine if it works and its safety.

The purpose of this research is to gather additional information on the safety and effectiveness of both Quetiapine and Pimavanserin. By doing this study, the investigators hope to learn which of these medications is the most effective course of treatment for people with PD psychosis.

Enrollment is open to Veterans nationwide, see your VA provider about the possibility of being referred to one of the study's Hub sites. This can be done through contact from your provider to the study's NSC (Tamara Boney at 267-303-9829).

DETAILED DESCRIPTION:
CSP #2015 - C-SAPP is a randomized, intent-to-treat, double-blind, two-arm, parallel design, multicenter comparator study. A total of up to approximately 24 Department of Veterans Affairs Medical Centers (VAMCs) will be invited to participate in the study. Veterans age 40 years and older with PD and symptoms of psychosis will be pre-screened for enrollment (consent) using established inclusion/exclusion criteria. Enrolled participants meeting eligibility will be randomized in a blinded fashion to one of two arms (fixed-dose pimavanserin or flexible-dose quetiapine), stratified by cognitive impairment [per the Montreal Cognitive Assessment (MoCA)]. Assessments will be collected at multiple time points - baseline, week 3, week 5, and at week 8 after randomization. Assessments of psychosis (CGI-I psychosis), PDP symptoms (SAPS-PD), and nighttime sleep/daytime sleepiness [per Scales for Outcomes in PD-Sleep Scale nighttime subscale (SCOPA-S NS)/Epworth Sleepiness Scale (ESS)] will be completed at each in-person visit, while caregiver burden (ZBI), functioning and well-being [per the Parkinson's Disease Questionnaire-8 (PDQ-8)] will be assessed at baseline and treatment visits of weeks 5 and 8, parkinsonism (CGI-I parkinsonism) and motor abilities (MDS-UPDRS III) at baseline and week 8, and cognition (MoCA) at screening and week 8. Additional contact by phone/video will occur at weeks 1 and 6. PD medications and side-effects will also be collected. SAEs, and AEs using the Treatment Emergent Symptom Scale (TESS) for guidance, will be continuously monitored at each participant contact (in-person and phone/video). A quality by design (QbD) approach was utilized focusing on its key principles to help prospectively identify important errors that could jeopardize the reliability of the data and safety of study participants.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Age 40 years or older
* Diagnosis of Parkinson's Disease consistent with UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria
* Psychosis [with Neuropsychiatric Inventory (NPI) hallucinations (B) or delusions (A) score 4 or greater]
* Stable dose of PD medications for at least 2 weeks
* If on an acetylcholinesterase inhibitor (AChEI) initially prescribed at least 3 months prior and stable dose (no dose or medication change) for past month
* Informed other must provide informed consent and agree to attend all study visits. The informed other must be at least 18 years of age and have regular contact with the patient (on average at least 4 days per week and at least 2 hours per day, or at least 3 days per week and at least 4 hours per day, that is with patient) via in-person, video, or telephone
* English-speaking

INFORMED OTHER

* Age 18 years or older
* Must have regular contact with the patient (on average at least 4 days per week, and at least 2 hours per day, or at least 3 days per week and at least 4 hours pr day, that is with patient) via in-person, video, or telephone
* Agree to attend all study visits
* Be able to provide informed consent
* English-speaking

Exclusion Criteria:

* Psychosis symptoms severe enough to preclude enrollment in a clinical trial and require prompt clinical care instead
* Treatment with quetiapine >50 mg/day or pimavanserin in the past 3 months, or quetiapine 50 mg/day or another antipsychotic in the past week prior to study randomization
* Deep brain stimulation (DBS) surgery within 3 months or has had stimulator adjustments in the previous 2 weeks
* History of a psychotic disorder prior to PD, including bipolar disorder, schizophrenia, schizoaffective disorder, and major depressive disorder with psychotic features, if it is thought to be the cause of the current psychosis symptoms
* Suspected atypical parkinsonian disorder or dementia with Lewy bodies (DLB)
* Psychosis secondary to other toxic or metabolic disorder
* History of long QT syndrome
* Documented chart evidence indicating persistent hypoglycemia, hypokalemia, hypomagnesemia that would put patient at increased risk for QTc prolongation.
* History of ventricular arrhythmias, except when treated with an implantable cardioverter defibrillator (ICD) or pacemaker, or untreated or unstable atrial fibrillation/flutter
* Currently taking medications that are moderate or strong CYP3A4 inducers or strong CYP3A4 inhibitors
* Concomitant use of drugs that prolong the QTc interval with a known risk of Torsades de Pointes
* Comorbid medical condition determined too severe by Site Investigator to allow participation in clinical trial
* Failure to tolerate quetiapine or pimavanserin previously
* Severe cognitive impairment (MoCA score <5)
* Nursing home placement at screening or planned placement during the study, unless approved by study Co-Chairs. Approval will depend upon nursing facility agreement to receive, return, and administer medications or allow participant to self-administer study medications; appropriate IO availability; and transportation availability for study visits.
* Currently enrolled in another therapeutic or interventional study
* Pregnant, or a female of child-bearing potential who is unwilling to use a reliable form of contraception

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2026-10-24 (Estimated); Study Completion 2027-08-24 (Estimated)

PRIMARY OUTCOMES:
CGI-I Psychosis | 8 Weeks
  The Clinical Global Impressions (CGI) scale is a brief, well-established research rating tool used to quantify and track patient progress and treatment response over time. The CGI comprises two measures, one of which is Improvement (CGI-I) from the initiation of treatment. It is scored 1 to 7. The CGI-I is used to assess how much the patient's illness has improved or worsened relative to baseline when the intervention was started (1-Very much improved, 2-Much improved, 3-Minimally improved, 4-No change, 5-Minimally worse, 6-Much worse, 7-Very much worse). The CGI-I can also be used to assess specific domains, including psychosis (this study's primary outcome) and parkinsonism (a secondary outcome). During the 8 weeks, the CGI-I (for psychosis, hereafter simply referred to as the CGI-I) will be administered to all participants at 3 weeks, 5 weeks, and 8 weeks following a CGI-I baseline interview to assess clinical improvement in psychosis.

SECONDARY OUTCOMES:
SAPS-PD | 8 Weeks
  The primary assessment of change in psychosis severity is the score on the 9-item Parkinson's disease Scale for Assessment of Positive Symptoms (SAPS-PD). The SAPS-PD scale will assess positive symptoms, including hallucinations, delusions, bizarre behavior, and positive formal thought disorder. A clinical interview is used to evaluate the participant's symptoms. Items include: 1 Auditory Hallucinations; 2 Voices Conversing; 3 Somatic or Tactile Hallucinations; 4 Visual Hallucinations; 5 Global Rating of Severity of Hallucinations; 6 Persecutory Delusions; 7 Delusions of Jealousy; 8 Ideas and Delusions of Reference; and 9 Global Rating of Severity of Delusions. Each item is given a score ranging 0 to 5 (0-None, 1-Questionable, 2-Mild, 3-Moderate, 4-Marked, 5-Severe). During the 8 weeks, the SAPS-PD will be administered to all participants at baseline, 3 weeks, 5 weeks, and 8 weeks to assess symptoms of PDP and psychopharmacological response to treatment.
MDS-UPDRS III | 8 Weeks
  The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (Motor Examination; MDS-UPDRS III) has 33 scores across 18 items (each score 0-4, range of total score 0-132, with higher scores indicating more severe motor symptoms) is completed by a trained rater during an examination of the patient, and is the most commonly-used assessment of parkinsonism in clinical trials. MDS-UPDRS III includes ratings for tremor, slowness (bradykinesia), stiffness (rigidity), and gait/balance. The MDS-UPDRS III will be administered to all participants at baseline and 8 weeks.
CGI-I Parkinsonism | 8 Weeks
  The Clinical Global Impressions (CGI) scale is a brief, rating tool used to quantify and track patient progress and treatment response over time. It was developed to be used in clinical trials on mental health to provide an assessment of the clinician's view of the patient's global functioning over time with a study medication. The CGI comprises two measures, but the one to be used in this study is Improvement (CGI-I) from the st of treatment. It is scored from 1 to 7. The CGI-I is used to assess how much the patient's illness has improved or worsened relative to baseline when the intervention was started (1-Very much improved, 2-Much improved, 3-Minimally improved, 4-No change, 5-Minimally worse, 6-Much worse, 7-Very much worse). The CGI-I (for parkinsonism) will be administered to all participants at 8 weeks following a CGI-I baseline interview to assess improvement in parkinsonism.
Zarit Caregiver Burden Scale | 8 Weeks
  The Zarit Burden Interview (ZBI) is a 22-item self-report inventory that examines burden associated with functional/behavioral impairments and the home care situation. It was developed to measure subjective burden among caregivers of adults with dementia. The items are worded subjectively, focusing on the affective response of the caregiver. Each question is scored on a 5-point Likert scale ranging from 0 to 4 (0-Never, 1-Rarely, 2-Sometimes, 3-Frequently, 4-Nearly always). The ZBI total score ranges from 0 (low burden) to 88 (high burden), the sum of the scores from all 22 questions. Interpretation of the total scores is: 1) 0-21 little or no burden; 2) 21-40 mild to moderate burden; 3) 41-60 moderate to severe burden; and 4) 61-88 severe burden. The ZBI will be administered to all participants' informed other at baseline and treatment phase visits of Weeks 5 and 8.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weintraub, MD, Study Chair — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (24):
- United States (24):
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Lexington VA Medical Center, Lexington, KY, Lexington, Kentucky
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - Asheville VA Medical Center, Asheville, NC, Asheville, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Philadelphia MultiService Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No